CLINICAL TRIAL: NCT05349721
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel Study to Assess the Efficacy, Safety, Tolerability, PK, and Biomarker Effects of PTC857 in Adult Subjects With Amyotrophic Lateral Sclerosis (CARDINALS)
Brief Title: Study to Assess the Effects of PTC857 Treatment in Participants With Amyotrophic Lateral Sclerosis ALS
Acronym: CARDINALS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company decision
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTC857-CNS-001-ALS; 2021-006511-29 (EudraCT Number); 2023-510317-26-00 (Other: EU CT Number)
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Results first posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PTC857 (Experimental): Participants will receive PTC857 during the 24-Week Treatment Period.
  Following successful completion of the Treatment Period, participants who enter the Long-term Extension (LTE) Period, will receive open-label PTC857 for 28 weeks. Following completion of the LTE period, participants who enter the Continued LTE Period will receive open-label PTC857 for an additional 108 weeks.
  Interventions: Drug: PTC857
- Placebo (Active Comparator): Participants will receive matching placebo during the 24-Week Treatment Period.
  Following successful completion of the Treatment Period, participants who enter the LTE Period, will receive open-label PTC857 for 28 weeks. Following completion of the LTE period, participants who enter the Continued LTE Period will receive open-label PTC857 for an additional 108 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PTC857 — PTC8657 will be administered as an oral solution twice a day.
  Arms: PTC857
Drug: Placebo — Matching placebo will be administered as an oral solution twice a day.
  Arms: Placebo

SUMMARY:
This study will assess the efficacy and safety of PTC857 treatment in participants diagnosed with ALS.

DETAILED DESCRIPTION:
Participants will be randomized to 1 of the 2 treatment groups: PTC857 or matching placebo. Following successful completion of the Treatment Period, participants who enter the LTE Period, will receive open-label PTC857 for 28 weeks. Following completion of the LTE period, participants who enter the Continued LTE Period will receive open-label PTC857 for an additional 108 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* ALS with preserved function, defined as:

  1. Onset of the first symptom leading to the diagnosis of ALS ≤24 months at the time of the initial Screening Visit
  2. Revised EL Escorial criteria of either:

  (i) Clinically definite ALS (ii) Clinically probable ALS
* A total ALSFRS-R score of at least 34 at the start of the Screening Period
* No significant respiratory compromise as evidenced by slow vital capacity ≥60% at the start of the Screening Period
* All chronic concomitant medications (both prescription and over the counter), and non-pharmacologic therapy regimens, excluding standard-of-care therapy riluzole, edaravone, or sodium phenylbutyrate/taurursodiol, should be stable and unchanged from 14 days prior to the start of the Screening Period and intend to remain stable and unchanged throughout the course of the study
* Female participants must have a negative breast cancer imaging screening status (not considered clinically abnormal and/or requiring further evaluation/treatment) within 6 months prior to the Screening Visit, or during the Screening Period.
* Standard-of-care therapy for the treatment of ALS (riluzole, edaravone, or sodium phenylbutyrate/taurursodiol) should be stable and unchanged from 30 (-3) days prior to the start of the Screening Period and intend to remain stable and unchanged throughout the course of the study.

Key Exclusion Criteria:

* Females who are pregnant or nursing or plan to become pregnant during the study
* Participants with clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular/ischemic disease or any other condition that, in the opinion of the investigator would jeopardize the safety of the participant or impact the validity of the study results
* Any clinically significant medical or psychiatric condition or medical history that, in the opinion of the investigator or the medical monitor, would interfere with the participant's ability to participate in the study or increase the risk of participation for that participant
* Current participation in any other investigational study with an investigational product or participation within 30 days prior to the start of the Screening Period or 5 half-lives of the previously taken investigational drug, whichever is longer
* Participant has previously received PTC857
* Participant is receiving a combination of edaravone and sodium phenylbutyrate/taurursodiol treatment, where applicable, within 30 days prior to the start of the Screening Period
* For female participants, any past medical history of breast cancer, regardless of remission status, or any first degree relative with history of breast cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2024-09-26 (Actual); Study Completion 2025-01-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (55):
- United States (14):
  - UC Irvine Health ALS and Neuromuscular Center, Orange, California
  - Forbes Norris MDA/ALS Research Center at California Pacific Medical Center, San Francisco, California
  - Holy Cross Hospital, Phil Smith Neuroscience Institute, Fort Lauderdale, Florida
  - University of South Florida - Carol and Frank Morsani Center for Advanced Healthcare, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - University of Kansas Medical Center (KUMC) - Landon Center on Aging, Kansas City, Kansas
  - Henry Ford Health System Department of Neurology, Detroit, Michigan
  - Neurology Associates, P.C. / Somnos Clinical Research, Lincoln, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Providence Brain and Spine Institute, Portland, Oregon
  - Lewis Katz School of Medicine at Temple Universtiy, Philadelphia, Pennsylvania
  - National Neuromuscular Research Institute, Austin, Texas
  - Nerve and Muscle Center of Texas, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (3):
  - STAT Research S.A., Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Iadin Srl., Buenos Aires
  - Hospital Ramos Mejía, Buenos Aires
- Australia (4):
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Gold Coast Hospital, Southport, Queensland
  - Calvary Health Care Bethlehem, Caulfield South, Victoria
  - Austin Health, Heidelberg, Victoria
- Belgium (2):
  - AZ Sint-Lucas Gent, Ghent
  - UZ Leuven, Leuven
- Czechia (2):
  - University hospital Brno, Department of Neurology, Brno
  - FORBELI s.r.o., Prague
- France (7):
  - CHU de Bordeaux, Bordeaux
  - Hôpital Neurologique Pierre Wertheimer, Bron
  - CHU Gabriel Montpied, Clermont-Ferrand
  - CHRU Lille - Hôpital Roger Salengro, Lille
  - CHU Dupuytren 1 Limoges, Limoges
  - CHU Gui de Chauliac (Pharmacie Saint-Eloi & Gui de Chauliac, Hopital Saint-Eloi), Montpellier
  - CRMR SLA - MNM du CHU de Nice, Nice
- Germany (5):
  - Charite - Universitatsmedizin - Berlin, Berlin
  - Hannover Medical School, Hanover
  - University Hospital Jena, Jena
  - Universitaetsklinikum Schleswig-Holstein (UKSH) Campus Luebeck, Klinik fuer Neurologie, Praezisionsneurologie, Lübeck
  - University of Ulm, Dept. of Neurology, Ulm
- Italy (9):
  - Centro Clinico Nemo Brescia, Brescia
  - Istituti Clinici Scientifici Maugeri IRCCS, Milan
  - Istituto Auxolgoico Italiano, Milan
  - Azienda Ospedaliero Universitaria di Modena, Modena
  - Maggiore della Carita University Hospital, Neurology department, ALS center, Novara
  - ALS Clinical Research Center, University Hospital Policlinico "P Giaccone", Palermo
  - IRCCS Fondazione Mondino - Reparto Neuroncologia/Neuroinfiammazione, Pavia
  - Policlinico Umberto I, Roma
  - AOU Citta Della Salute e Scienza, Torino
- PTC Clinical Site, Japanese City, Japan
- UMC Utrecht, Utrecht, Netherlands
- Poland (2):
  - Centrum Medyczne Neuro Protect, Warsaw
  - City Clinic Research Sp. Z o.o, Warsaw
- Spain (3):
  - Unidad Neuromuscular. Servicio de Neurologia Hospital Universitari Vall d'Hebron, Barcelona
  - H. St Pau, Barcelona
  - Hospital Universitario y Politecnico La Fe, Valencia
- Sweden (2):
  - Skanes universitetssjukhus, VE Neurologi, Malmo
  - Norrlands universitetssjukhus Neurologens Forskningsavdelning, Umeå

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included Treatment (Part A), long-term extension (LTE) (Part B), and Continued LTE (Part C) periods.
Groups:
- Utreloxastat: Participants received utreloxastat during the 24-Week Treatment Period. Following successful completion of the Treatment Period, participants who entered the LTE Period received open-label utreloxastat for 28 weeks. Following completion of the LTE period, participants who entered the Continued LTE Period received open-label utreloxastat for an additional 108 weeks.
- Placebo: Participants received matching placebo during the 24-Week Treatment Period. Following successful completion of the Treatment Period, participants who entered the LTE Period received open-label utreloxastat for 28 weeks. Following completion of the LTE period, participants who entered the Continued LTE Period received open-label utreloxastat for an additional 108 weeks.
Period: Part A (24 Weeks)
Arm/Group | Utreloxastat | Placebo
Started | 222 | 114
Received at Least 1 Dose of Double-blind Study Drug in the Part A | 220 | 114
Completed | 179 | 100
Not Completed | 43 | 14
Not completed — Adverse Event | 9 | 2
Not completed — Death | 8 | 3
Not completed — Disease Progression | 1 | 1
Not completed — Screen Failure | 2 | 0
Not completed — Withdrawal by Subject | 18 | 7
Not completed — Other Than Specified | 5 | 1
Period: Part B (28 Weeks)
Arm/Group | Utreloxastat | Placebo
Started | 173 | 100
Received at Least 1 Dose of Open-label Utreloxastat During Part B | 173 | 100
Completed | 38 | 27
Not Completed | 135 | 73
Not completed — Adverse Event | 3 | 0
Not completed — Death | 21 | 11
Not completed — Disease Progression | 2 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Study terminated by sponsor | 85 | 53
Not completed — Withdrawal by Subject | 17 | 5
Not completed — Other Than Specified | 4 | 2
Period: Part C (108 Weeks)
Arm/Group | Utreloxastat | Placebo
Started | 35 | 27
Received at Least 1 Dose of Open-label Utreloxastat During Part C | 35 | 27
Completed | 0 | 1
Not Completed | 35 | 26
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Study terminated by sponsor | 34 | 23
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety set included all randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Utreloxastat | Placebo | Total
Number analyzed (Participants) | 220 | 114 | 334
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (10.97) | 57.1 (9.88) | 57.7 (10.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 28 | 105
  Male | 143 | 86 | 229
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 19 | 46
  Not Hispanic or Latino | 189 | 93 | 282
  Unknown or Not Reported | 4 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 183 | 96 | 279
  Race: Black or African Descent | 5 | 0 | 5
  Race: Asian Descent | 10 | 5 | 15
  Race: Other | 22 | 13 | 35

OUTCOME MEASURES:

1. Primary Outcome: Combined Assessment of Function (ALS Functional Rating Scale-Revised [ALSFRS-R]) and Survival (CAFS) Rank After 24 Weeks of Treatment (Intention-to-Treat [ITT] 1 Analysis Population)
Description: The CAFS is a composite endpoint based on time to earlier occurrence of death and change from baseline in ALSFRS-R score. ALSFRS-R is a rating scale where 12 functions were rated on 5-point scales (from 0 to 4) with a maximum score of 48 (sum of all 12 items), with a higher score indicating better function. Each participant's outcome was compared to every other participant's outcome in a pairwise fashion by time to death and change on ALSFRS-R, assigned a score which was sum of comparisons (+1 [better], 0 [tie], -1 [worse]), and summed scores were ranked, from 1 to 306 (ITT1 Analysis Set) lowest rank corresponds to participant who died first and highest rank to the participant with best ALSFRS-R outcome among those who survived. Multiple imputation was used to impute participants with missing ALSFRS-R score at Week 24. A higher rank was considered a better outcome. Least square (LS) means and standard error (SE) were calculated using analysis of covariance (ANCOVA) model.
Time Frame: Week 24
Population: ITT1 Analysis Set included all randomized participants who received at least 1 dose of double-blind study drug in the Treatment Period and who had a decrease in the ALSFRS-R score of ≤4 points during the Screening Period.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Utreloxastat | Placebo
Number analyzed (Participants) | 202 | 104
units on a scale | 172.22 (13.25) | 165.36 (14.65)
Statistical Analysis 1: Comparison: Utreloxastat vs Placebo; Test type: Other; p = 0.516, ANCOVA; Estimates were derived from the ANCOVA model (following multiple imputation), where participant ranks served as the response variable; Treatment Difference = 6.86, 95% CI 2-sided [-13.86 to 27.59]

2. Secondary Outcome: Combined Assessment of Function (ALSFRS-R) and Survival (CAFS) Rank After 24 Weeks of Treatment (ITT2 Analysis Population)
Description: The CAFS is a composite endpoint based on time to earlier occurrence of death and change from baseline in ALSFRS-R score. ALSFRS-R is a rating scale where 12 functions were rated on 5-point scales (from 0 to 4) with a maximum score of 48 (sum of all 12 items), with a higher score indicating better function. Each participant's outcome was compared to every other participant's outcome in a pairwise fashion by time to death and change on ALSFRS-R, assigned a score which was sum of comparisons (+1 [better], 0 [tie], -1 [worse]), and summed scores were ranked, from 1 to 334 (ITT2 Analysis Set) lowest rank corresponds to participant who died first and highest rank to the participant with best ALSFRS-R outcome among those who survived. A higher rank was considered a better outcome. LS mean and SE were calculated using ANCOVA model.
Time Frame: Week 24
Population: ITT2 Analysis Set included all randomized participants who received at least 1 dose of double-blind study drug in the Treatment Period.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Utreloxastat | Placebo
Number analyzed (Participants) | 220 | 114
units on a scale | 188.58 (14.81) | 181.89 (15.96)

3. Secondary Outcome: Change From Baseline in ALSFRS-R Score at Week 24 (ITT1 Analysis Population)
Description: The ALSFRS-R is a quickly administered (5-minute) ordinal rating scale that assesses the participant's capability and independence in 12 functional activities across 4 subdomains of bodily function (bulbar, gross motor, fine motor, and respiratory) relevant in ALS. Each activity was recorded to the closest approximation from a list of 5 choices, scored 0 (total loss of function) to 4 (no loss of function), with the total score ranging from 0 to 48 and higher scores indicating less functional impairment. LS mean and SE were calculated using mixed model repeated measures (MMRM).
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Utreloxastat | Placebo
Number analyzed (Participants) | 202 | 104
units on a scale | 29.4 (0.73) | 31.4 (0.93)

4. Secondary Outcome: Change From Baseline in ALSFRS-R Score at Week 24 (ITT2 Analysis Population)
Description: The ALSFRS-R is a quickly administered (5-minute) ordinal rating scale that assesses the participant's capability and independence in 12 functional activities across 4 subdomains of bodily function (bulbar, gross motor, fine motor, and respiratory) relevant in ALS. Each activity was recorded to the closest approximation from a list of 5 choices, scored 0 (total loss of function) to 4 (no loss of function), with the total score ranging from 0 to 48 and higher scores indicating less functional impairment. LS mean and SE were calculated using MMRM.
Time Frame: Baseline, Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Utreloxastat | Placebo
Number analyzed (Participants) | 220 | 114
units on a scale | 27.7 (0.71) | 29.1 (0.88)

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and non-serious AEs. A TEAE was defined as an AE that began after the first administration of study drug or any existing AEs that worsened after the first dose of study drug. A summary of other non-serious AEs and all SAEs, regardless of causality is located in the 'Reported AE section'.
Time Frame: Day 1 through Week 24
Population: Safety set included all randomized participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Utreloxastat | Placebo
Number analyzed (Participants) | 220 | 114
Participants | 174 | 90

6. Secondary Outcome: Change From Baseline in Percent Predicted Slow Vital Capacity (SVC) at Week 24
Description: The SVC is a measure of breathing function. SVC measures the volume that can be exhaled from a full inhalation after exhaling to a maximum as slowly as possible. The percent of predicted SVC is reported. LS mean and SE were calculated using MMRM.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent predicted SVC
Arm/Group | Utreloxastat | Placebo
Number analyzed (Participants) | 202 | 104
percent predicted SVC | -14.62 (2.106) | -15.92 (2.518)

7. Secondary Outcome: Change From Baseline in Modified Norris Scale Total Score at Week 24
Description: Modified Norris scale is used to assess the motor/limb and bulbar function. The Modified Norris Scale is a rating scale for ALS that consists of 2 parts: the Limb Norris Scale and the Norris Bulbar Scale. The Limb Norris Scale has 21 items to evaluate extremity function, and the Norris Bulbar Scale has 13 items to evaluate bulbar function. Each item was rated in 4 ordinal categories, corresponding to the following values and ratings or functional scores: normal (3 points), somewhat impaired (2 points), inadequate (1 point), and "cannot do at all" (0 points). The total score was calculated by summing all the scales, ranging from 0 (worst) to 102 (best) where higher scores indicated better functional abilities. LS mean and SE were calculated using MMRM.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Utreloxastat | Placebo
Number analyzed (Participants) | 202 | 104
units on a scale | -18.2 (1.57) | -18.0 (1.82)

8. Secondary Outcome: Overall Survival Rate
Description: Overall survival rate was defined as percentage of participants who were alive at given timepoint. Overall survival was defined as the time in months from the date of first dose to the date of death from any cause or date last known alive for those who did not die.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Utreloxastat | Placebo
Number analyzed (Participants) | 202 | 104
percentage of participants | 95.8 [92.9 to 98.6] | 97.9 [95.1 to 100.0]

9. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time in months from the date of first dose to the date of death from any cause or date last known alive for those who did not die.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Utreloxastat | Placebo
Number analyzed (Participants) | 202 | 104
months | NA [NA to NA] — Due to smaller number of participants with an event, median and 95% confidence interval (CI) could not be calculated. | NA [NA to NA] — Due to smaller number of participants with an event, median and 95% CI could not be calculated.

10. Secondary Outcome: Change From Baseline in ALS Assessment Questionnaire (ALSAQ-40) Total Score at Week 24
Description: The ALSAQ-40 is a disease-specific measure of health-related quality of life (QOL) for ALS. The ALSAQ-40 is comprised of 40 questions measuring 5 discrete dimensions of health status that are affected by the disease: physical mobility (10 items); activities of daily living and independence (10 items); eating and drinking (3 items); communication (7 items); emotional reactions (10 items). Participants were asked to indicate the frequency of each event by selecting one of 5 options (Likert scale: 0-4): never/rarely/sometimes/often/ always or cannot do at all. The total score ranging from 0 (no impairment) to 160 (severe impairment) was calculated by adding the 5 domain scores. A lower score indicates a better health state. LS mean and SE were calculated using MMRM.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Utreloxastat | Placebo
Number analyzed (Participants) | 202 | 104
units on a scale | 27.9 (3.05) | 23.9 (3.48)

11. Secondary Outcome: Change From Baseline in Neurofilament Light Chain (NfL) Activity at Week 24
Description: The NfL is a marker of axonal degeneration and is robustly elevated in the blood of many neurological and neurodegenerative conditions.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Geometric Mean (Standard Error); unit: picograms (pg)/milliliter (mL)
Arm/Group | Utreloxastat | Placebo
Number analyzed (Participants) | 202 | 104
picograms (pg)/milliliter (mL) | 69.98 (6.69) | 64.75 (7.08)

12. Secondary Outcome: Area Under the Concentration-time Curve From 0 to Measurable Timepoint (AUC0-t) of Utreloxastat in Plasma
Time Frame: Day 1 and Day 29
Population: Pharmacokinetic (PK) analysis set included all randomized participants who received at least 1 dose of double-blind study drug in the Treatment Period and had at least 1 measurable post-baseline plasma or CSF utreloxastat concentration. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: hours*nanograms (ng)/mL
Arm/Group | Utreloxastat
Number analyzed (Participants) | 13
hours*nanograms (ng)/mL
  Day 1 | 2670 (1330)
  Day 29: number analyzed (Participants) | 12
  Day 29 | 4220 (1110)

13. Secondary Outcome: Maximum Observed Concentration (Cmax) of Utreloxastat in Plasma
Time Frame: Day 1 and Day 29
Population: PK analysis set included all randomized participants who received at least 1 dose of double-blind study drug in the Treatment Period and had at least 1 measurable post-baseline plasma or CSF utreloxastat concentration. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Utreloxastat
Number analyzed (Participants) | 13
ng/mL
  Day 1 | 796 (492)
  Day 29: number analyzed (Participants) | 12
  Day 29 | 881 (397)

14. Secondary Outcome: Mean Concentration of Utreloxastat in Cerebrospinal Fluid (CSF)
Time Frame: Day 1 and Day 29
Population: PK analysis set included all randomized participants who received at least 1 dose of double-blind study drug in the Treatment Period and had at least 1 measurable post-baseline plasma or CSF utreloxastat concentration. 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Utreloxastat
Number analyzed (Participants) | 9
ng/mL
  Day 1 | NA (NA) — Data not estimable due to below limit of quantification (BLQ).
  Day 29: number analyzed (Participants) | 8
  Day 29 | NA (NA) — Data not estimable due to BLQ.

ADVERSE EVENTS:
Time Frame: Day 1 through Week 141
Description: Part A: Safety set included all randomized participants who received at least 1 dose of study drug.
  Part B and C: Long-term extension safety set included all participants who received at least 1 dose of the open-label study drug during the long-term extension periods.
  Per pre-specified, the long-term extension AE data was collected and reported combined for Part B and Part C.
Groups:
- Part A: Utreloxastat: Participants received utreloxastat during the 24-Week Treatment Period.
- Part A: Placebo: Participants received matching placebo during the 24-Week Treatment Period.
- Parts B and C: Utreloxastat/Utreloxastat; Parts B and C: Placebo/ Utreloxastat: Following successful completion of the Treatment Period, participants who entered the LTE Period received open-label utreloxastat for 28 weeks. Following completion of the LTE period, participants who entered the Continued LTE Period received open-label utreloxastat for an additional 108 weeks.
Arm/Group | Part A: Utreloxastat | Part A: Placebo | Parts B and C: Utreloxastat/Utreloxastat | Parts B and C: Placebo/ Utreloxastat
All-Cause Mortality (participants affected / at risk) | 9/220 | 3/114 | 23/173 | 15/100
Serious Adverse Events (participants affected / at risk) | 36/220 | 11/114 | 48/173 | 25/100
Other Adverse Events (participants affected / at risk) | 167/220 | 88/114 | 115/173 | 53/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Utreloxastat (N=220) | Part A: Placebo (N=114) | Parts B and C: Utreloxastat/Utreloxastat (N=173) | Parts B and C: Placebo/ Utreloxastat (N=100)
Pneumonia (Infections and infestations) | 4 | 0 | 7 | 3
Respiratory tract infection (Infections and infestations) | 3 | 0 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 1 | 1 | 2 | 0
Abscess (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia pneumococcal (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 12 | 10
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 5 | 0
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 3
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0 | 2
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 3 | 1
Autoimmune pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Death (General disorders) | 1 | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 1 | 2 | 3
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0
Coronavirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Device related sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Hypercapnic coma (Nervous system disorders) | 0 | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Euthanasia (Surgical and medical procedures) | 0 | 0 | 1 | 0
Jejunostomy (Surgical and medical procedures) | 0 | 0 | 0 | 1
Otolithiasis (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Troponin increased (Investigations) | 0 | 0 | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Device dislocation (Product Issues) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Utreloxastat (N=220) | Part A: Placebo (N=114) | Parts B and C: Utreloxastat/Utreloxastat (N=173) | Parts B and C: Placebo/ Utreloxastat (N=100)
Diarrhoea (Gastrointestinal disorders) | 21 | 17 | 6 | 5
Nausea (Gastrointestinal disorders) | 17 | 9 | 7 | 0
Constipation (Gastrointestinal disorders) | 11 | 6 | 9 | 3
Vomiting (Gastrointestinal disorders) | 9 | 2 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 7 | 3 | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 3 | 3 | 0
Flatulence (Gastrointestinal disorders) | 3 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 2 | 0
Oral discomfort (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 2 | 0
Aerophagia (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Angular cheilitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal hypermotility (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Leukoplakia oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Mucous stools (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Tongue discolouration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Tooth discolouration (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 4 | 1 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 4 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 7 | 11 | 2 | 2
COVID-19 (Infections and infestations) | 11 | 5 | 10 | 2
Urinary tract infection (Infections and infestations) | 12 | 1 | 8 | 2
Influenza (Infections and infestations) | 5 | 4 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 3 | 5 | 1
Gastroenteritis (Infections and infestations) | 6 | 0 | 2 | 0
Respiratory tract infection (Infections and infestations) | 4 | 2 | 1 | 2
Oral candidiasis (Infections and infestations) | 3 | 2 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 3 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 3 | 1 | 2 | 1
Sinusitis (Infections and infestations) | 3 | 1 | 1 | 0
Pharyngitis (Infections and infestations) | 2 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 1 | 0
Coronavirus infection (Infections and infestations) | 2 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 1 | 1 | 0 | 1
Oral herpes (Infections and infestations) | 2 | 0 | 0 | 1
Tinea pedis (Infections and infestations) | 1 | 1 | 0 | 0
Abscess (Infections and infestations) | 1 | 0 | 0 | 0
Asymptomatic bacteriuria (Infections and infestations) | 1 | 0 | 0 | 0
Catheter site infection (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0
Mumps (Infections and infestations) | 1 | 0 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 1 | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 2 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0 | 0 | 0
Stoma site infection (Infections and infestations) | 1 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0
Tracheitis (Infections and infestations) | 0 | 1 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 36 | 17 | 30 | 12
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 8 | 2 | 2 | 0
Skin laceration (Injury, poisoning and procedural complications) | 5 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 4 | 1 | 2 | 0
Head injury (Injury, poisoning and procedural complications) | 3 | 1 | 3 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 2 | 1 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 3 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Chillblains (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lip injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Nasal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post procedural complication circulatory (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 29 | 14 | 8 | 2
Dizziness (Nervous system disorders) | 5 | 4 | 2 | 0
Presyncope (Nervous system disorders) | 3 | 1 | 1 | 0
Syncope (Nervous system disorders) | 2 | 2 | 1 | 0
Taste disorder (Nervous system disorders) | 3 | 1 | 0 | 0
Ageusia (Nervous system disorders) | 2 | 1 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 2 | 1 | 1 | 0
Sciatica (Nervous system disorders) | 2 | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 2 | 0 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 0 | 2 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 0 | 1 | 1 | 0
Meralgia paraesthetica (Nervous system disorders) | 0 | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Muscle spasticity (Nervous system disorders) | 1 | 0 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 1 | 0 | 0 | 0
Transient global amnesia (Nervous system disorders) | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 4 | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 3 | 4 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 2 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 1 | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Shoulder girdle pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 18 | 7 | 2 | 0
Pyrexia (General disorders) | 6 | 1 | 7 | 2
Asthenia (General disorders) | 4 | 0 | 0 | 1
Oedema peripheral (General disorders) | 3 | 1 | 3 | 1
Peripheral swelling (General disorders) | 3 | 0 | 0 | 0
Chills (General disorders) | 1 | 1 | 0 | 0
Pain (General disorders) | 2 | 0 | 0 | 0
Catheter site bruise (General disorders) | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0
Crying (General disorders) | 0 | 1 | 0 | 0
Gait inability (General disorders) | 0 | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0
Hyperthermia (General disorders) | 1 | 0 | 0 | 0
Illness (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 1 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Oedema (General disorders) | 1 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 1 | 5 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Paranasal sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 9 | 4 | 3 | 0
Anxiety (Psychiatric disorders) | 3 | 2 | 1 | 1
Depression (Psychiatric disorders) | 3 | 2 | 3 | 0
Sleep disorder (Psychiatric disorders) | 4 | 0 | 3 | 0
Suicidal ideation (Psychiatric disorders) | 3 | 1 | 0 | 0
Mood altered (Psychiatric disorders) | 3 | 0 | 2 | 0
Adjustment disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Affective disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 1 | 0 | 1 | 0
Claustrophobia (Psychiatric disorders) | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 1 | 1 | 0
Libido increased (Psychiatric disorders) | 1 | 0 | 0 | 0
Mixed anxiety and depressive disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 9 | 3 | 6 | 2
Hypotension (Vascular disorders) | 2 | 4 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 0 | 2 | 1
Hot flush (Vascular disorders) | 1 | 2 | 0 | 0
Haematoma (Vascular disorders) | 2 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0 | 0
Aortic arteriosclerosis (Vascular disorders) | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0
White coat hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 3 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 3 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 3 | 0 | 3 | 1
Blood pressure increased (Investigations) | 2 | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 2 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 2 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 4 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 4 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 1 | 0
Blood magnesium decreased (Investigations) | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 1 | 0
Full blood count abnormal (Investigations) | 1 | 0 | 0 | 0
Liver function test increased (Investigations) | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 1
Mean cell volume increased (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 6 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 3 | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypozincaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 1 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 0 | 2 | 0
Polyuria (Renal and urinary disorders) | 1 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 2 | 0 | 0 | 0
Renal cyst (Renal and urinary disorders) | 2 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0
Bladder disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Neurogenic bladder (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urge incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary tract inflammation (Renal and urinary disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 3 | 3 | 1 | 0
Palpitations (Cardiac disorders) | 2 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 5 | 0 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0
Anaemia macrocytic (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 4 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 2 | 0 | 1 | 1
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Motion sickness (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 2 | 1 | 0 | 0
Eye irritation (Eye disorders) | 1 | 1 | 0 | 0
Vision blurred (Eye disorders) | 2 | 0 | 0 | 0
Conjunctival irritation (Eye disorders) | 0 | 1 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 1 | 0 | 0
Eyelid ptosis (Eye disorders) | 1 | 0 | 0 | 0
Hepatic cyst (Hepatobiliary disorders) | 2 | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Nipple pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Type V hyperlipidaemia (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Colostomy (Surgical and medical procedures) | 0 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 1
Helicobacter infection (Infections and infestations) | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Lyme disease (Infections and infestations) | 0 | 0 | 1 | 0
Nasal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Bone contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Stoma site pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Tongue coated (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Burning sensation (Nervous system disorders) | 0 | 0 | 1 | 0
Hypotonia (Nervous system disorders) | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 1 | 0
Discomfort (General disorders) | 0 | 0 | 1 | 0
Granuloma (General disorders) | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 1 | 0
Swelling face (General disorders) | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory muscle weakness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 1
Breath sounds abnormal (Investigations) | 0 | 0 | 1 | 0
Cardiac murmur (Investigations) | 0 | 0 | 1 | 0
Differential white blood cell count abnormal (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram ST-T change (Investigations) | 0 | 0 | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 0 | 1 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 1 | 0
Respiratory rate increased (Investigations) | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 1 | 0
Ultrasound breast abnormal (Investigations) | 0 | 0 | 1 | 0
Urine analysis abnormal (Investigations) | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0
Behaviour disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Enuresis (Psychiatric disorders) | 0 | 0 | 1 | 0
Pallor (Vascular disorders) | 0 | 0 | 1 | 0
Post thrombotic syndrome (Vascular disorders) | 0 | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Lividity (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Macrocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Crystalluria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Cardiac dysfunction (Cardiac disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 0 | 1 | 0
Chalazion (Eye disorders) | 0 | 0 | 0 | 1
Eyelid myokymia (Eye disorders) | 0 | 0 | 1 | 0
Contrast media allergy (Immune system disorders) | 0 | 0 | 1 | 0
Immunisation reaction (Immune system disorders) | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cardiac septal defect (Congenital, familial and genetic disorders) | 0 | 0 | 1 | 0
Gastrostomy (Surgical and medical procedures) | 0 | 0 | 1 | 0
Secretion discharge (General disorders) | 1 | 0 | 0 | 0
Pharyngitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early due to company decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review results and/or communications prior to public release and can embargo communications regarding trial results for a period that is up to 180 days from the time submitted to the sponsor for review. The sponsor may consult with the PI to require changes to the communication or extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2024-06-14): https://cdn.clinicaltrials.gov/large-docs/21/NCT05349721/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-25): https://cdn.clinicaltrials.gov/large-docs/21/NCT05349721/SAP_001.pdf